CLINICAL TRIAL: NCT02479386
Title: A Multicenter, Prospective Epidemiologic Study of The Progression of Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: A Study of Disease Progression in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Acronym: Proxima A
Status: Terminated | Type: Observational
Why Stopped: There is no longer a plan to pursue an approval of lampalizumab.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: GX29633; 2014-003939-19 (EudraCT Number); GX29639 (Other: Hoffmann-La Roche ID)
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

GROUPS / COHORTS (1):
- Cohort Geographic Atrophy: Cohort of participants with GA secondary to AMD will be evaluated for changes in GA over time.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was administered in this study.

SUMMARY:
This study seeks to better characterize relationships between visual function and the progression (worsening) of geographic atrophy (GA) due to age-related macular degeneration (AMD). The study is also intended to generate new information on the relationship between genetics and GA progression. This is a global, prospective, multicenter, epidemiologic study enrolling participants with GA secondary to AMD. The study visits are scheduled to occur every 6 months. The anticipated duration of the study is up to 48 months. There is a planned interim analysis around the 2-year time window for the study.

ELIGIBILITY:
Inclusion Criteria:

* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year for at least 30 days after the last fluorescein dye administration
* The study is being conducted in participants with GA in both Study Eye and Non-Study Eye (bilateral GA) with no evidence of prior or active choroidal neovascularization (CNV)

Exclusion Criteria:

* Previous participation in any studies of investigational drugs for GA or dry AMD (except for studies of vitamins and minerals)
* GA in either eye due to causes other than AMD
* History of vitrectomy surgery, submacular surgery, or any surgical intervention for AMD
* Previous laser photocoagulation for CNV, diabetic macular edema, retinal vein occlusion, and/or proliferative diabetic retinopathy
* Any ocular or systemic medical conditions that, in the opinion of the investigator, could contribute to participant's inability to participate in the study or interfere with study assessments
* Requirement for continuous use of therapy indicated in Prohibited Therapy in the study Protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Scotomatous Points as Assessed by Mesopic Microperimetry (MP) | Baseline up to end of study (up to approximately 48 months)
Macular Sensitivity as Assessed by Mesopic MP | Baseline up to end of study (up to approximately 48 months)
Best Corrected Visual Acuity (BCVA) Score as Assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart | Baseline up to end of study (up to approximately 48 months)
BCVA Score as Assessed by ETDRS Chart Under Low Luminance Conditions | Baseline up to end of study (up to approximately 48 months)
Monocular and Binocular Reading Speed as Assessed by the Minnesota Low-Vision Reading Test (MNRead) or by Radner Reading Cards | Baseline up to end of study (up to approximately 48 months)
Monocular and Binocular Critical Print Size as Assessed by the MNRead or by Radner Reading Cards | Baseline up to end of study (up to approximately 48 months)

SECONDARY OUTCOMES:
Change from Baseline in the GA area, as Assessed by Fundus Autofluorescence (FAF) | Baseline, end of study (up to approximately 48 months)
Change from Baseline in National Eye Institute Visual Functioning Questionnaire 25-item Version (NEI VFQ-25) Score | Baseline, end of study (up to approximately 48 months)
Change from Baseline in Functional Reading Independence (FRI) Index Score | Baseline, end of study (up to approximately 48 months)
Percentage of Participants With Medical Events of Interest (MEIs) | Baseline up to end of study (up to approximately 48 months)
  The clinical events (cardiovascular, respiratory, cognitive, ocular events etc.) occurring during the study are termed as MEIs. These events will be collected using MEI electronic Case Report Form (eCRF) checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (91):
- United States (23):
  - Northwest Arkansas Retina Associates, Springdale, Arkansas
  - Retinal Diagnostic Center, Campbell, California
  - Specialty Eye Care Medical Center, Glendale, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - East Bay Retina Consultants, Oakland, California
  - Colorado Retina Associates, PC, Golden, Colorado
  - Rand Eye, Deerfield Beach, Florida
  - Bascom Palmer Eye Institute, Naples, Florida
  - Center For Sight, Sarasota, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Paducah Retinal Center, Paducah, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Foundation for Vision Research, Grand Rapids, Michigan
  - MaculaCare, PLLC, New York, New York
  - Vitreous-Retina-Macula, New York, New York
  - University of North Carolina; Kittner Eye Center, Chapel Hill, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Duke University Eye Center; Vitreoretinal, Durham, North Carolina
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Palmetto Retina Center, Florence, South Carolina
  - Retina Consultants of Houston, Houston, Texas
  - Med Center Ophthalmology Assoc, San Antonio, Texas
  - Wagner Macula & Retina Center, Norfolk, Virginia
- Argentina (6):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Oftalmos, Capital Federal
  - Centro Privado de Ojos Romagosa, Córdoba
  - Onnis Instituto oftalmológico privado, Córdoba
  - Clinica Privada de Ojos, Mar del Plata
  - Centro Oftalmólogos Especialistas, Rosario
- Australia (5):
  - Northern Beaches Retina Cataract Glaucoma, Mona Vale, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Newcastle Eye Hospital Research Foundation, Waratah, New South Wales
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Medizinische Universität Wien; Universitätsklinik für Augenheilkunde und Optometrie, Vienna, Austria
- Brazil (5):
  - Hospital de Olhos de Aparecida - HOA, Aparecida de Goiânia, Goiás
  - Instituto da Visão, Belo Horizonte, Minas Gerais
  - Botelho Hospital da Visao, Blumenau, Santa Catarina
  - Instituto da Visão IPEPO, São Paulo, São Paulo
  - Hosp Clinicas da FMUSP, São Paulo, São Paulo
- Canada (2):
  - Calgary Retina Consultants, Calgary, Alberta
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
- France (10):
  - Chi De Creteil; Ophtalmologie, Créteil
  - Clinique de la Louviere - Nord retine; Maladie et chirurgie des Yeux, Lille
  - Centre ophtalmologique Rabelais; Ophtalmologie, Lyon
  - Centre Paradis Monticelli; Ophtalmologie, Marseille
  - Hopital Lariboisiere; Ophtalmologie, Paris
  - CHNO des Quinze Vingts; Ophtalmologie, Paris
  - Fondation Rothschild; Ophtalmologie, Paris
  - CHU Poitiers - CHR La Miletrie; Ophtalmologie, Poitiers
  - Centres Ophtalmologique St Exupéry; Ophtalmologie, Saint-Cyr-sur-Loire
  - Cabinet La Maison Rouge; Ophtalmologie, Strasbourg
- Germany (3):
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar der TU München; Augenklinik, München
  - Universitätsklinikum Tübingen, Tübingen
- Greece (2):
  - University General Hospital of Heraklion; Department of Ophthalmology, Heraklion
  - European Interbalkan Medical Center; Ophthalmology Dpt, Thessaloniki
- Hungary (4):
  - Bajcsy-Zsilinszky Hospital, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont; Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest
  - Kenezy Gyula Korhaz; Szemeszet, Debrecen
  - Markusovszky Egyetemi Oktatokorhaz ; SZEMESZET, Szombathely
- Israel (8):
  - Soroka university medical center; Ophtalmology, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah MC; Ophtalmology, Jerusalem
  - Meir Medical Center; Ophtalmology, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center; Ophtalmology, Rehovot
  - Tel Aviv Sourasky MC; Ophtalmology, Tel Aviv
- Italy (6):
  - Università degli Studi di Napoli Federico II; Dipartimento di Scienze Oftalmologiche, Napoli, Campania
  - ASST FATEBENEFRATELLI SACCO; Oculistica (Sacco), Milan, Lombardy
  - Università degli Studi dell'Insubria; Clinica Oculistica, Varese, Lombardy
  - Azienda Ospedaliero-Universitaria Careggi; S.O.D. Oculistica, Florence, Tuscany
  - Nuovo Ospedale S. Chiara - A.O.U.P Presidio Ospedaliero di Cisanello; U.O. Oculistica Universitaria, Pisa, Tuscany
  - Ospedale Classificato Equiparato Sacro Cuore - Don Calabria; Dipartimento Oculistica, Negrar - Verona, Veneto
- Poland (3):
  - Klinika Okulistyki Ogolnej w Lublinie, Lublin
  - Pomorski Uniwersytet Medyczny w Szczecinie, Zaklad Patologii Ogolnej PUM", Szczecin
  - SPEKTRUM Osrodek Okulistyki Klinicznej, Wroclaw
- Spain (6):
  - Institut de la Macula i la retina, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oftalmologia, Barcelona
  - Hospital Universitario Virgen de la Macarena; Servicio de Oftalmologia, Seville
  - Clinica Doctores Piñero; Oftalmologia, Seville
  - Hospital Clinico Universitario de Valladolid; Servicio de oftalmologia, Valladolid
  - Hospital Universitario Rio Hortega; Servicio de Oftalmologia, Valladolid
- United Kingdom (7):
  - Bristol Eye Hospital, Bristol
  - Kent & Canterbury Hospital, Canterbury
  - Hull and East Yorkshire Eye Hospital, Hull
  - John Radcliffe Hospital; Oxford Eye Hospital, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southhampton
  - Sunderland Eye Infirmary, Sunderland
  - Pinderfields Hospital; Clinical Research Team, Rowan House, Wakefield

REFERENCES:
- [Derived] Salvi A, Cluceru J, Gao SS, Rabe C, Schiffman C, Yang Q, Lee AY, Keane PA, Sadda SR, Holz FG, Ferrara D, Anegondi N. Deep Learning to Predict the Future Growth of Geographic Atrophy from Fundus Autofluorescence. Ophthalmol Sci. 2024 Oct 23;5(2):100635. doi: 10.1016/j.xops.2024.100635. eCollection 2025 Mar-Apr. PMID 39758130
- [Derived] Anegondi N, Steffen V, Sadda SR, Schmitz-Valckenberg S, Tufail A, Csaky K, Lad EM, Kaiser PK, Ferrara D, Chakravarthy U. Visual Loss in Geographic Atrophy: Learnings from the Lampalizumab Trials. Ophthalmology. 2025 Apr;132(4):420-430. doi: 10.1016/j.ophtha.2024.11.017. Epub 2024 Nov 23. PMID 39581330
- [Derived] Cluceru J, Anegondi N, Gao SS, Lee AY, Lad EM, Chakravarthy U, Yang Q, Steffen V, Friesenhahn M, Rabe C, Ferrara D. Topographic Clinical Insights From Deep Learning-Based Geographic Atrophy Progression Prediction. Transl Vis Sci Technol. 2024 Aug 1;13(8):6. doi: 10.1167/tvst.13.8.6. PMID 39102242
- [Derived] Spaide T, Jiang J, Patil J, Anegondi N, Steffen V, Kawczynski MG, Newton EM, Rabe C, Gao SS, Lee AY, Holz FG, Sadda S, Schmitz-Valckenberg S, Ferrara D. Geographic Atrophy Segmentation Using Multimodal Deep Learning. Transl Vis Sci Technol. 2023 Jul 3;12(7):10. doi: 10.1167/tvst.12.7.10. PMID 37428131